CLINICAL TRIAL: NCT03657524
Title: Combined Thoracic Ultrasound Using Speckle Tracking for the Prediction of Weaning Failure : a Prospective Multicenter Study
Brief Title: Speckle Tracking Echocardiography for the Prediction of Weaning Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-34
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Weaning Failure of Mechanical Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resuscitation patients (Experimental)
  Interventions: Other: echocardiography
- healthy volunteers (Active Comparator)
  Interventions: Other: echocardiography

INTERVENTIONS:
Other: echocardiography — Speckle tracking echocardiography

SUMMARY:
Deciding the optimal timing for extubation in patients who are mechanically ventilated can be challenging, and traditional weaning predictor tools are not accurate. Recent studies suggest that isolated sonographic assessment of the respiratory and cardiac function (ie diastolic function and filling pressure), in mechanically ventilated patients may assist in identifying patients at risk of weaning failure. Recently, the association of conventional echocardiography and lung ultrasound showed promising results for the prediction of post extubation distress. Speckle Tracking is an emerging tool in intensive care medicine that has never been investiguated for the prediction of weaning failure. It could early detects diastolic dysfunction and and elevated filling pressure. Of more, speckle tracking is known to be less operator dependant. The main objective of our study is to evaluate the diagnosis accuracy of speckle tracking echocardiography performed during a weaning trial to predict weaning failure. The secondary objectives are to assess the diagnosis accuracy of combined heart and lung ultrasound to predict weaning failure.

DETAILED DESCRIPTION:
Deciding the optimal timing for extubation in patients who are mechanically ventilated can be challenging, and traditional weaning predictor tools are not accurate. Recent studies suggest that isolated sonographic assessment of the respiratory and cardiac function (ie diastolic function and filling pressure), in mechanically ventilated patients may assist in identifying patients at risk of weaning failure. Recently, the association of conventional echocardiography and lung ultrasound showed promising results for the prediction of post extubation distress. Speckle Tracking is an emerging tool in intensive care medicine that has never been investiguated for the prediction of weaning failure. It could early detects diastolic dysfunction and and elevated filling pressure. Of more, speckle tracking is known to be less operator dependant. The main objective of our study is to evaluate the diagnosis accuracy of speckle tracking echocardiography performed during a weaning trial to predict weaning failure. The secondary objectives are to assess the diagnosis accuracy of combined heart and lung ultrasound to predict weaning failure.

ELIGIBILITY:
Inclusion Criteria:

- Patients hospitalized in intensive care unit under mechanical fulfilling the criteria of ventilation weaning trial.

Exclusion Criteria:

* Less than 18 years old.
* Pregnancy
* Non sinusal cardiac rhythm
* Neuro Myopathy
* Tracheotomy
* Lack of echogenicity to perform at least a four chamber apical view

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2026-05-21 (Estimated); Study Completion 2026-05-21 (Estimated)

PRIMARY OUTCOMES:
lung and heart ultrasounds | Just before and during the weaning trial
  Area under the receiver operator characteristic curve (AUC) of global longitudinal strain and strain rate variations (before and during a weaning trial) to predict weaning failure.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France